CLINICAL TRIAL: NCT02101125
Title: A Phase 1 Open-label, Single-sequence Study to Evaluate the Effect of Concomitant Administration of BMS-986020 on the Single-dose Pharmacokinetics of Rosuvastatin in Healthy Subjects
Brief Title: Drug Interaction Study With Rosuvastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None
Other Study IDs: IM136-122
Record Dates: First submitted 2014-03-28; First posted 2014-04-01 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-06

CONDITIONS: Immunosuppression For Disease
MeSH Terms: interventions — lysophosphatidic acid; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BMS-986020 + Rosuvastatin (Treatment A, B and C) (Experimental): Cohort 1: Rosuvastatin Tablet Single dose and BMS- 986020 orally on specific days
  Cohort 2 (Administered 4 hrs, after the morning dose of BMS-986020): Rosuvastatin Tablet Single dose and BMS- 986020 orally on specific days
  Interventions: Drug: BMS-986020; Drug: Rosuvastatin

INTERVENTIONS:
Drug: BMS-986020
  Other Names: Lysophosphatidic acid (LPA1) Antagonist
Drug: Rosuvastatin
  Other Names: Crestor

SUMMARY:
The purpose of this study is to evaluate the effect of concomitant administration of BMS-986020 on the single dose Pharmacokinetics (PK) of Rosuvastatin in healthy subjects.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Healthy subjects who have no clinically significant deviation from normal in medical history, surgical history, PE, vital signs, ECG, and clinical laboratory determinations
* Nonsmokers
* Body Mass Index (BMI) of 18.0 to 32.0 kg/m2, inclusive. Men, ages 18 to 50 years, inclusive
* Men and women, ages 18 to 50 years, inclusive
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of investigational product
* Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug(s) (11 days) plus 5 half-lives of the study drug (4 days) plus 90 days (duration of sperm turnover) for a total of 94 days posttreatment completion

Exclusion Criteria:

* Any significant acute or chronic medical illness
* Current or recent (within 3 months of study drug administration) gastrointestinal disease
* Any major surgery within 4 weeks of study drug administration
* Any gastrointestinal surgery (eg, partial gastrectomy, pyloroplasty) including cholecystectomy that could impact upon the absorption of study drug
* Donation of > 400 mL of blood within 8 weeks or donation of plasma (except at screening visit) within 4 weeks of study drug administration
* Blood transfusion within 4 weeks of study drug administration
* Inability to tolerate oral medication
* Inability to be venipunctured and/or tolerate venous access as determined by the investigator
* Use of tobacco-containing or nicotine containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patches, nicotine lozenges, or nicotine gum) within 6 months prior to check-in, or a positive nicotine test (ie, cotinine) at screening or check-in
* Subjects who drink more than 3 cups of coffee or other caffeine containing products with an equivalent amount of caffeine per day, or 5 cups of tea per day
* History of allergy to Lysophosphatidic acid (LPA1) antagonists or related compounds

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2014-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of Rosuvastatin with and without coadministered BMS-986020 | 31 timepoints up to Day 12
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration (AUC(0-T)) of Rosuvastatin with and without coadministered BMS-986020 | 31 timepoints up to Day 12
Area under the plasma concentration-time curve from time zero extrapolated to infinite time (AUC(INF)) of Rosuvastatin with and without coadministered BMS-986020 | 31 timepoints up to Day 12

SECONDARY OUTCOMES:
Time of maximum observed plasma concentration (Tmax) of Rosuvastatin with and without coadministered BMS-986020 | 31 timepoints up to Day 12
Terminal plasma half-life (T-HALF) of Rosuvastatin with and without coadministered BMS-986020 | 31 timepoints up to Day 12
Apparent total body clearance (CLT/F) of Rosuvastatin with and without coadministered BMS-986020 | 31 timepoints up to Day 12
Incidence of Adverse Event (AEs), Serious Adverse Event (SAEs), deaths, and AEs leading to discontinuation | Upto Day 12
Results of vital signs, ECGs, Physical Examination (PEs), and clinical lab result | Up to Day 12

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Healthcare Discoveries, Llc D/B/A Icon Development Solutions, San Antonio, Texas, United States

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx